CLINICAL TRIAL: NCT00715676
Title: A Phase 2, Double-blind, Randomized, Placebo-Controlled, Daily-dose, Proof-of-concept Study of a Vitamin D Compound in Postmenopausal Women With Osteopenia
Brief Title: Phase 2 Safety and Efficacy Study of a Vitamin D Compound (DP001) in Postmenopausal Women With Low Bone Mineral Density
Acronym: 2MD-3H-2B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deltanoid Pharmaceuticals (Industry)
Responsible Party: Hector F. DeLuca, President and Chief Executive Officer, Deltanoid Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Deltanoid 2MD-3H-2B
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2009-12

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; 2-methylene-19-nor-(20S)-1a, 25-dihydroxyvitamin D3; Vitamin D; Bone Density Conservation Agents; Bone Regeneration
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Group 2 (Experimental): 220 ng
  Interventions: Drug: DP001
- Group 3 (Experimental): 440 ng
  Interventions: Drug: DP001

INTERVENTIONS:
Drug: Placebo — oral, once daily
  Arms: Group 1
Drug: DP001 — oral, once daily
  Other Names: 2-methylene-19-nor-(20S)-1a, 25-dihydroxyvitamin D3; 2MD
  Arms: Group 2; Group 3

SUMMARY:
This study will evaluate the effect of a 1-year administration of the vitamin D analog 2-methylene-19-nor-(20S)-1alpha, 25-dihydroxyvitamin D3 (DP001) on bone mineral density (BMD), safety, and tolerability.

DETAILED DESCRIPTION:
DP001 is a vitamin D analog that has been shown to stimulate bone formation in pre-clinical studies. In a Phase 1B study of postmenopausal women, an increase in the bone formation marker, osteocalcin, was evident without an increase in serum calcium. The aim of this study is to determine if 1-year administration of DP001 to postmenopausal women with osteopenia results in a significant increase in BMD at doses that are safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female subjects, defined as amenorrheic for at least 5 years
* Body Mass Index of 18 to 35
* Osteopenic
* Generally healthy
* Informed consent

Exclusion Criteria

* History or evidence of acute or unstable chronic hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, psychiatric, or neurologic diseases
* Current or recent treatment with any medications or products affecting vitamin D metabolism, calcium balance, bone turnover, or an investigational drug therapy
* 12-lead electrocardiogram demonstrating QTc (QT interval corrected for heart rate) >450 milliseconds at screening
* Abnormal creatinine clearance
* Elevated urinary calcium levels
* Vitamin D deficiency
* Excessive dietary calcium or vitamin D intake
* Current use of any illicit drug and/or history of alcohol abuse

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A Bedale, Ph.D., Study Director — Deltanoid Pharmaceuticals
Locations (9):
- United States (9):
  - Boling Clinical Trials, Upland, California
  - Indiana School of Medicine University Hospital, Indianapolis, Indiana
  - Bethesda Health Research, Bethesda, Maryland
  - Creighton University Bone Metabolism Unit, Omaha, Nebraska
  - New Mexico Clinical Research and Osteoporosis Center, Albuquerque, New Mexico
  - Winthrop University Hospital Bone Mineral Research Center, Mineola, New York
  - Helen Hayes Hospital Clinical Research Center, West Haverstraw, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Wisconsin-Madison Osteoporosis Clinical Research, Madison, Wisconsin

REFERENCES:
- [Background] Ke HZ, Qi H, Crawford DT, Simmons HA, Xu G, Li M, Plum L, Clagett-Dame M, DeLuca HF, Thompson DD, Brown TA. A new vitamin D analog, 2MD, restores trabecular and cortical bone mass and strength in ovariectomized rats with established osteopenia. J Bone Miner Res. 2005 Oct;20(10):1742-55. doi: 10.1359/JBMR.050605. Epub 2005 Jun 13. PMID 16160732
- [Background] Plum LA, Fitzpatrick LA, Ma X, Binkley NC, Zella JB, Clagett-Dame M, DeLuca HF. 2MD, a new anabolic agent for osteoporosis treatment. Osteoporos Int. 2006;17(5):704-15. doi: 10.1007/s00198-005-0036-3. Epub 2006 Feb 21. PMID 16491322
- [Background] Shevde NK, Plum LA, Clagett-Dame M, Yamamoto H, Pike JW, DeLuca HF. A potent analog of 1alpha,25-dihydroxyvitamin D3 selectively induces bone formation. Proc Natl Acad Sci U S A. 2002 Oct 15;99(21):13487-91. doi: 10.1073/pnas.202471299. Epub 2002 Oct 8. PMID 12374862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 5 March 2007 to 19 December 2007 at 9 centers within the United States.
Groups:
- Placebo: Placebo soft gel capsules, oral, once daily
- 220 ng of Vitamin D Analog (DP001): 220 ng DP001 soft gel capsules, oral, once daily DP001 is also known as 2-methylene-19-nor-(20S)-1alpha, 25-dihydroxyvitamin D3.
- 440 ng DP001: 440 ng DP001 soft gel capsules, oral, once daily
Period: Overall Study
Arm/Group | Placebo | 220 ng of Vitamin D Analog (DP001) | 440 ng DP001
Started | 49 (1 additional subject was enrolled in the placebo group but discontinued before taking any study drug) | 54 | 53
Completed | 43 | 43 | 21
Not Completed | 6 | 11 | 32
Not completed — Adverse Event | 3 | 5 | 21
Not completed — Withdrawal by Subject | 1 | 3 | 8
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Terminated by Sponsor | 1 | 0 | 0
Not completed — Did Not Meet Entry Criteria | 0 | 0 | 1
Not completed — Use of Exclusionary Medication | 0 | 0 | 1
Not completed — Elevated Blood Glucose | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 220 ng DP001: 220 ng DP001 soft gel capsules, oral, once daily
- Total: Total of all reporting groups
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001 | Total
Number analyzed (Participants) | 49 | 54 | 53 | 156
Age Continuous [Mean (Standard Deviation); unit: years] | 61.1 (6.5) | 61.6 (5.5) | 61.9 (5.3) | 61.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 53 | 156
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Week 52
Description: Percent change in lumbar spine BMD (relative to baseline) at Week 52
Time Frame: Baseline and Week 52
Population: This analysis was performed on the Full Analysis Set, which included all subjects who received at least one dose of study drug. Multiple imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Number analyzed (Participants) | 49 | 54 | 53
Percent change | -0.537 (2.545) | -0.174 (2.820) | 0.309 (3.904)
Statistical Analysis 1: Comparison: Placebo vs 220 ng DP001; A sample size of 49 per treatment group was calculated to have at least 90% power to detect a 2% or greater increase over placebo assuming the following: (1) a standard deviation of the percent change of 2.75% (2) a dropout rate of 30%, and (3) one-sided 0.05 level of significance; Test type: Superiority or Other; p = 0.641, ANOVA — The Hochberg method was used to compare dose groups to placebo and control the Type 1 error rate
Statistical Analysis 2: Comparison: Placebo vs 440 ng DP001; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.243, ANOVA — The Hochberg method was used to compare dose groups to placebo and control the Type 1 error rate

2. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 52
Description: The percent change in hip BMD (relative to baseline) at Week 52
Time Frame: Baseline and Week 52
Population: This analysis was conducted on the Full Analysis Set, which included all randomized subjects who received at least one dose of study drug. Multiple imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Number analyzed (Participants) | 49 | 54 | 53
Percent Change | -0.315 (1.894) | -0.540 (1.782) | -0.887 (1.833)
Statistical Analysis 1: Comparison: Placebo vs 220 ng DP001; Test type: Superiority or Other; p = 0.778, ANOVA
Statistical Analysis 2: Comparison: Placebo vs 440 ng DP001; Test type: Superiority or Other; p = 0.173, ANOVA

3. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density (BMD) at Week 52
Description: Percent change in femoral neck BMD (relative to baseline) at Week 52
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Number analyzed (Participants) | 49 | 54 | 53
Percent change | -0.428 (2.511) | -1.085 (3.150) | -0.680 (2.507)
Statistical Analysis 1: Comparison: Placebo vs 220 ng DP001; Test type: Superiority or Other; p = 0.395, ANOVA
Statistical Analysis 2: Comparison: Placebo vs 440 ng DP001; Test type: Superiority or Other; p = 0.523, ANOVA

4. Secondary Outcome: Percent Change From Baseline in Trochanter Bone Mineral Density (BMD) at Week 52
Description: Percent change in trochanter BMD (relative to baseline) at Week 52
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Number analyzed (Participants) | 49 | 54 | 53
Percent change | -0.375 (2.604) | -0.341 (2.565) | -0.941 (2.554)
Statistical Analysis 1: Comparison: Placebo vs 220 ng DP001; Test type: Superiority or Other; p = 0.928, ANOVA
Statistical Analysis 2: Comparison: Placebo vs 440 ng DP001; Test type: Superiority or Other; p = 0.124, ANOVA

5. Secondary Outcome: Change From Baseline in Serum Calcium Levels at Week 52
Description: Change in serum calcium value (relative to baseline) at Week 52
Time Frame: Baseline and Week 52
Population: This analysis was done for all subjects for whom both baseline and Week 52 data was available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Number analyzed (Participants) | 43 | 43 | 21
mg/dL | -0.06 (0.268) | 0.11 (0.286) | 0.29 (0.243)
Statistical Analysis 1: Comparison: Placebo vs 220 ng DP001; Test type: Superiority or Other; Mean Difference (Net) = 0.173, 90% CI [0.164 to 0.181]
Statistical Analysis 2: Comparison: Placebo vs 440 ng DP001; Test type: Superiority or Other; Mean Difference (Net) = 0.582, 90% CI [0.573 to 0.591]

6. Secondary Outcome: Percent Change From Baseline in Serum Bone Markers at Week 26
Description: Percent change from baseline at Week 26
Time Frame: Baseline and Week 26
Population: Analyses were performed using subjects for whom both Baseline and Week 26 samples were available.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Number analyzed (Participants) | 45 | 45 | 29
Percent change
  Serum C-telopeptide cross-links of type 1 collagen | 4.5 (25.4) | 13.8 (32.4) | 54.5 (54.2)
  Osteocalcin | 3.8 (19.4) | 22.4 (38.0) | 80.3 (73.3)
  Procollagen type 1 N-propeptide | 1.0 (29.5) | 11.8 (40.7) | 9.2 (33.4)

7. Secondary Outcome: Number of Subjects With at Least 1 Treatment-emergent Adverse Event
Description: To assess safety and tolerability, the number of subjects in each treatment group who had one or more adverse events recorded after the beginning of study drug administration were determined.
Time Frame: 1 year
Population: The participants for this analysis included all randomized subjects who received a dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Number analyzed (Participants) | 49 | 54 | 53
Participants | 41 | 45 | 46

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a period of 1 year for subjects completing the study, and through study discontinuation for subjects who discontinued early.
Description: Adverse events were assessed by investigator assessment at subject visits and regular laboratory testing.
Arm/Group | Placebo | 220 ng DP001 | 440 ng DP001
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/54 | 3/53
Other Adverse Events (participants affected / at risk) | 38/49 | 37/54 | 44/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | 220 ng DP001 (N=54) | 440 ng DP001 (N=53)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | 220 ng DP001 (N=54) | 440 ng DP001 (N=53)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 8
Blood creatinine increased (Investigations) | 0 | 1 | 4
Bronchitis (Infections and infestations) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 5 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 4
Fatigue (General disorders) | 1 | 3 | 6
Gastroenteritis viral (Infections and infestations) | 3 | 1 | 1
Headache (Nervous system disorders) | 4 | 7 | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 13
Hypercalciuria (Renal and urinary disorders) | 0 | 7 | 12
Hypertension (Vascular disorders) | 4 | 1 | 1
Influenza (Infections and infestations) | 4 | 1 | 4
Insomnia (Psychiatric disorders) | 2 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Nasopharyngitis (Infections and infestations) | 10 | 11 | 6
Nausea (Gastrointestinal disorders) | 5 | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3
Pyrexia (General disorders) | 3 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 3 | 1
Stomach discomfort (Gastrointestinal disorders) | 4 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 4
Urinary tract infection (Infections and infestations) | 5 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days